CLINICAL TRIAL: NCT05462899
Title: Purpose in Life, Goals, and Expectations of Older Adults After Hospitalization and Their Caregivers
Brief Title: Purpose in Life, Goals, and Expectations
Status: Not yet recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Maureen C. Ashe, Principal Investigator, University of British Columbia
Other Study IDs: H21-03607
Record Dates: First submitted 2022-07-11; First posted 2022-07-18 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Goals

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Purpose in life, goals, and expectations — There is no intervention. This is a cross-sectional study.

SUMMARY:
Study investigators are inviting participants to participate in a study to describe older adults' and family caregivers' purpose in life, goals, and expectations for recovery after hospitalization. Study investigators will ask older adults and caregivers to take part in a telephone or online interview to ask questions and answer questionnaires related to their experience with the hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Older adults 60y+ and family caregivers
* after hospitalization

Exclusion Criteria:

* We will exclude older adults with a dementia diagnosis, head injury, significant neurological impairment, not expected to live for 6 months or longer, or who receive treatment for medical conditions precluding enrolment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Older adults 60y+ and family caregivers after hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Experience and perceptions after hospitalization | 1 day
  Semi-structured interviews

SECONDARY OUTCOMES:
Falls Efficacy Scale-International (FES-I) | 1 day
  A measure of a person's concern about falling. There are 16 items, each scored on a Likert scale with 1=not concerned and 4=very concerned. Higher scores indicate higher concerns fro falling.
Community Healthy Activities Model Program for Seniors (CHAMPS) Questionnaire | 1 day
  Physical activity questionaire which records the frequency and duration of a person's activities
Life-Space questionnaire | 1 day
  A measure of a person's mobility within their home, neighbourhood, and beyond (e.g., spatial movement). Participants respond yes/no to where they have been within the past 3 days (e..g., home, outside home in the neighborhood, etc.
Functional Independence Measure | 1 day
  A measure of disability with a focus on self-care, transfers, walking, communication, and social cognition. It is an 18-item (7-level) ordinal scale. For each item (scored 1-7), the higher the score the more dependent the person is on the task.
Occupational Balance Questionnaire (Short form) | 1 day
  Records the satisfaction with the amount and variation of a person's activities. It has 11 items with 4-step ordinal scales. Higher scores indicate higher occupational balance.
Telephone Interview for Cognitive Status (TICS) to screen for cognitive impairment | 1 day
  A brief assessment of cognition for the telephone. There are 11 items, and the items are summed for a total TICS score. Results compared with previous dat at-scores and described qualitatively:Unimpaired, Ambiguous, Mildly Impaired, and Moderately to Severely Impaired
Hospital Anxiety and Depression Scale (HADS) | 1 day
  Measures anxiety and depression in patients. There are 7 questions each for anxiety and depression. The lower the number indicate less anxiety/depression. For example, a score less than 7 is considered a "non-case". Scores range from 0-21.
Ryff Scales of Psychological Well-Being | 1 day
  A 42-item scale which measures autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance. There are 42 statements using a 7-point scale (1 = strongly agree; 7 = strongly disagree). For overall score (all questions), higher scores suggest higher well-being.
EQ5D-5L | 1 day
  A self-reported health related quality of life measure. There are 5 categories and the person chooses their responses based on categories, from no problems to extreme problems for each category (mobility, self-care, usual activities, pain, anxiety/depression. An index score is created out of 1; a higher index score the better. participants would also rate their health (0-100) with 100 as the best possible health. The higher the score the
ICECAP-O | 1 day
  A self reported capability and well-being measure, with 5 attributes: attachment, security, role, enjoyment, and control. Index values out of 1, a higher value indicates higher reported capability and well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen C Ashe, PhD, Principal Investigator — UBC
Locations (1):
- The University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No